CLINICAL TRIAL: NCT06815692
Title: Effect of Interdisciplinary Interventions After Mild Traumatic Brain Injury
Brief Title: Interdisciplinary Interventions After mTBI
Status: Not yet recruiting | Type: Observational
Sponsor: Rune Skovgaard Rasmussen (Other)
Collaborators: Special Education and Employment Unit (SuB) in Slagelse, part of the municipality's Center for Disability and Psychiatry (Unknown); Danish Center for Concussion (Unknown)
Responsible Party: Sponsor-Investigator, Rune Skovgaard Rasmussen, MSc, Ph.D., associate professor, University Hospital, Gentofte, Copenhagen
Organization: University Hospital, Gentofte, Copenhagen (Other)
Other Study IDs: 12292024
Record Dates: First submitted 2025-01-23; First posted 2025-02-07 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Concussion, Mild
Keywords: mTBI; employment; weekly working hours; quality of life; Concussion
MeSH Terms: conditions — Brain Concussion | interventions — Physical Therapy Modalities; Restraint, Physical; Educational Status; Mindfulness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Early intervention: Interventions for mTBI patients initiated within 1 to 3 months after symptoms onset:
  Interventions include psychoeducation for the individual, their family, and their workplace or educational setting. Investigators initiate contact with the individual's workplace or educational setting to discuss the case and collaborate closely with both the individual and their employer/supervisor. Investigators focus on vocational rehabilitation, aiming to gradually increase the participant's work capacity, weekly working hours, and job retention. Ongoing supportive conversations are provided before and during work or study. Investigators offer counseling on cognitive and psychological aspects, with a focus on mental health.
  All interventions focus on gradual progression, exposure, and rehabilitation in both personal and work life. Participants are guided in gradually increasing activities and working hours.
  Interventions: Behavioral: Psychoeducation; Behavioral: Physiotherapy; Behavioral: Treatment of tinnitus and increased sound sensitivity; Behavioral: Vision training and examination; Behavioral: Sleep guidance and education; Behavioral: Mindfulness with a cognitive therapeutic approach; Behavioral: Employment-oriented intervention; Behavioral: Energy management and graded exercise; Other: Neuropsychological counseling
- Late intervention: Interventions for mTBI patients initiated at least 9 months after symptoms onset. Note that these interventions are the same as offered to the early interventions group:
  Interventions include psychoeducation for the individual, their family, and their workplace or educational setting. Investigators initiate contact with the individual's workplace or educational setting to discuss the case and collaborate closely with both the individual and their employer/supervisor. Investigators focus on vocational rehabilitation, aiming to gradually increase the participant's work capacity, weekly working hours, and job retention. Ongoing supportive conversations are provided before and during work or study. Investigators offer counseling on cognitive and psychological aspects, with a focus on mental health.
  All interventions focus on gradual progression, exposure, and rehabilitation in both personal and work life. Participants are guided in gradually increasing activities and working hours.
  Interventions: Behavioral: Psychoeducation; Behavioral: Physiotherapy; Behavioral: Treatment of tinnitus and increased sound sensitivity; Behavioral: Vision training and examination; Behavioral: Sleep guidance and education; Behavioral: Mindfulness with a cognitive therapeutic approach; Behavioral: Employment-oriented intervention; Behavioral: Energy management and graded exercise; Other: Neuropsychological counseling

INTERVENTIONS:
Behavioral: Psychoeducation — Focus on understanding mechanisms of concussion
Behavioral: Physiotherapy — Gradual training and physical exercises
Behavioral: Treatment of tinnitus and increased sound sensitivity — Treatment given individually or in groups
Behavioral: Vision training and examination — Training and examination by a neuro-optometrist
Behavioral: Sleep guidance and education — Counselling to achieve better sleep and reduce fatigue.
Behavioral: Mindfulness with a cognitive therapeutic approach — Training by certified mindfulness instructor
Behavioral: Employment-oriented intervention — The Concussion Team therapists work with a patient's employer to facilitate a gradual return to normal working hours.
Behavioral: Energy management and graded exercise — Counselling to achieve more energy and vitality.
Other: Neuropsychological counseling — Talks with a neuropsychologist about mTBI sequelae.

SUMMARY:
The investigators aim to investigate the impact of interdisciplinary and individually tailored programs for mTBI (concussion) on quality of life and work capacity, both at the conclusion of the program and after 1 and 3 years. The investigators also want to examine whether early intervention is significant by comparing individuals who enter the program between 1 and 3 months post-concussion with those who only start the program more than 9 months post-concussion. Such a study has not been conducted before and can provide valuable insights into long-term effects and the importance of early intervention

DETAILED DESCRIPTION:
A concussion typically results from a trauma to the head or body and, for most people, causes symptoms that resolve within a few weeks. Approximately 25,000 individuals in Denmark experience concussions annually. However, about 8,000 to 11,000 of those affected experience prolonged symptoms such as fatigue, dizziness, headaches, pain, and cognitive impairments. These symptoms can significantly reduce quality of life and work capacity, and in some cases, become chronic. Consequently, a subset of individuals with concussions require ongoing social support even two years post-injury.

Denmark currently lacks a comprehensive national guideline for managing concussions within regional and municipal healthcare systems. As a result, individuals with concussions are often left to navigate the healthcare system on their own, leading to limited or no access to rehabilitation services. The Danish Center for Concussion and other experts have recommended the establishment of national concussion clinics.

Since 2016, the Special Education and Employment Unit (SuB) in Slagelse, part of the municipality's Center for Disability and Psychiatry, has been developing and providing concussion interventions based on national and international evidence. Participants in these programs have reported significant improvements in weekly work hours and overall quality of life. However, the long-term effects of these interventions remain unknown.

Participants are typically in great distress and need help, which is why a lack of interventions-or the delay of interventions for several months-in a control group is considered unethical. It should be noted that single-group studies, which evaluate outcomes longitudinally, are often the only possible method and can provide both interesting and reliable results. Investigators will be blinded for participants being allocated to early or late interventions.

This single-center and uncontrolled study aims to investigate the long-term impact of interdisciplinary and personalized concussion rehabilitation programs on quality of life and work capacity. Researchers will compare the outcomes of individuals who begin the program within 1-3 months post-concussion to those who start later (more than 9 months post-concussion) to determine the significance of early intervention. This research is groundbreaking as it will provide valuable insights into the long-term effects of concussions and the importance of timely interventions.

Aim: To evaluate the effectiveness of tailored concussion rehabilitation programs.

Outcomes: Changes in quality of life and work capacity. Timeframes: Immediate post-program and at 1 and 3 years. Comparison: Early vs. late intervention. Significance: The study will fill a gap in the current understanding of concussion recovery.

In essence, this study seeks to determine if a comprehensive and individualized approach to concussion rehabilitation can lead to sustained improvements in the lives of those affected, and whether starting treatment sooner is beneficial.

The investigators expect that an early intervention will result in significantly higher average weekly work hours and quality of life compared to a late intervention. The main hypothesis is that an early intervention will counteract the chronic effects and prevent worsening, including by inhibiting the development of hypersensitivity to sound and light.

The vision is to offer an intervention for concussion sufferers at the highest international level, and with this focus, it is important to know the long-term effects.

ELIGIBILITY:
Inclusion Criteria:

* Adults who are medically diagnosed with a concussion.
* Adults with a connection to the labor market.
* Participants must be able to communicate in Danish and be able to independently participate in the intervention.
* Participants must be able to transport themsleves to and from SuB facility for their treatment sessions.
* Rivermead Post-Concussion Symptoms Questionnaire (RPQ) score must be at least 20, indicating a significant severity of symptoms following a concussion.

Exclusion Criteria:

* Persons without medically verified concussion.
* Person where brain injury was found at symptom onset.
* Persons with significant cognitive dysfunction.
* Persons who are unable to understand Danish or with communication disorders that hinder test performance.
* Persons with terminal illness or other progressive disease.
* Chronic use of opioids.
* Significant abuse of alcohol or euphoriants or narcotics or other serious illnesses that may affect test results or ability/possibility of attendance.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Two cohorts will be followed, one group of adults included between 1 and 3 months after a concussion, and another group experiencing a concussion 9 months before inclusion.
Sampling Method: Non-Probability Sample
Enrollment: 140 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2030-07-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Weekly working hours | Measured at inclusion, through study completion (an average of 6 months), and after 6, 12 and 36 months of no intervention
  Weekly working hours, measured in hours, will be assessed at baseline and after the intervention is completed. Subsequently, working hours will be assessed 1, 2, and 3 years after the intervention is completed. Follow-up will be conducted via telephone calls

SECONDARY OUTCOMES:
Rivermead Post-Concussion Symptoms Questionnaire (RPQ) | Measured at inclusion, through study completion (an average of 6 months), and after 6, 12 and 36 months of no intervention
  Scores range from 0 to 64, low scores are best.
Work Role Functioning Questionnaire v. 2.0 (WRFQ 2.0). | Measured at inclusion, through study completion (an average of 6 months), and after 6, 12 and 36 months of no intervention
  A higher score on the WRFQ 2.0 indicates better work role functioning. Scores range from 0 to 100.
Behavioural Rating Inventory of Executive Function - Adults (BRIEF-A) | Measured at inclusion, through study completion (an average of 6 months), and after 6, 12 and 36 months of no intervention
  T-scores are measured, a score above 65 indicates problems. Scores range from 0 to 99.
European Quality of Life - 5 Dimensions | Measured at inclusion, through study completion (an average of 6 months), and after 6, 12 and 36 months of no intervention
  Scores range from 0 to 100, high scores are best.
Clinical Global Impression Scale (CGI) | Measured at inclusion, through study completion (an average of 6 months), and after 6, 12 and 36 months of no intervention
  Scores range from 1 to 7, high score is worst.
Brain Injury Vision Symptom Survey (BIVSS) | Measured at inclusion, through study completion (an average of 6 months), and after 6, 12 and 36 months of no intervention
  The total score can range from 0 to 112. A higher score indicates a greater severity of visual symptoms.
King-Devick (K-D) | Measured at inclusion, through study completion (an average of 6 months), and after 6, 12 and 36 months of no intervention
  There is no strict range with clear cut-offs, normative data suggests that healthy individuals complete the test in under 60 seconds.
Vestibular Ocular Motor Screening (VOMS) | Measured at inclusion, through study completion (an average of 6 months), and after 6, 12 and 36 months of no intervention
  If symptoms are provoked, the individual rates their severity on a scale of 0 to 10 (0 = none, 10 = severe).
Reading test | Measured at inclusion, through study completion (an average of 6 months), and after 6, 12 and 36 months of no intervention
  Reading of a short article published in a newspaper. Faster reading times are best.
Major Depression Inventory (MDI) | Measured at inclusion, through study completion (an average of 6 months), and after 6, 12 and 36 months of no intervention
  Scores range from 0 to 50, low scores are best.
Fatigue Severity Scale - 7 item (FSS-7) | Measured at inclusion, through study completion (an average of 6 months), and after 6, 12 and 36 months of no intervention
  Scores range from 1 to 7. Low scores are best.
Visual Analogue Scale for Smerte (VAS) | Measured at inclusion, through study completion (an average of 6 months), and after 6, 12 and 36 months of no intervention
  Scores range from 0 to 10. Low scores are best.
Questionnaire about sound sensitivity and tinnitus | Measured at inclusion, through study completion (an average of 6 months), and after 6, 12 and 36 months of no intervention
  Scores range from 0 to 25, low scores are best.
Depression, Anxiety and Stress Scale (DASS42) | Measured at inclusion, through study completion (an average of 6 months), and after 6, 12 and 36 months of no intervention
  Scores range from 0 to 42, low scores are best.
Harvard Trauma Questionnaire (HTQ) | Measured at inclusion, through study completion (an average of 6 months), and after 6, 12 and 36 months of no intervention
  Scores ranged from 16 to 64. Low scores are best.
Generalized Anxiety Disorder Scale - 7 item (GAD-7) | Measured at inclusion, through study completion (an average of 6 months), and after 6, 12 and 36 months of no intervention
  Scores range from 0 to 21, low scores are best.

CONTACTS AND LOCATIONS:
Overall Officials: Rune S Rasmussen, MSc, PhD, Study Director — Special Education and Employment Unit (SuB) in Slagelse; Signe E Petersson, OT, Study Chair — Special Education and Employment Unit (SuB) in Slagelse

IPD SHARING:
Plan to Share IPD: No